CLINICAL TRIAL: NCT00818493
Title: An Open-Label Pilot Study of the Analgesic Efficacy and Safety Of Q8003 and of the Conversion From IV Morphine PCA Analgesia to Q8003 or to Percocet® in Patients Who Have Undergone Primary Unilateral Total Knee Arthroplasty or Total Hip Arthroplasty
Brief Title: Pilot Study of the Efficacy and Safety of Q8003 in Patients Who Have Undergone Total Knee Arthroplasty or Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: QRxPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q8003-020
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Postoperative Pain
Keywords: total knee arthroplasty; total hip arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — MoxDuo; Morphine; Oxycodone; oxycodone-acetaminophen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Q8003, flexible ascending dose
  Interventions: Drug: Q8003 (morphine sulfate and oxycodone hydrochloride)
- 2 (Experimental): Low dose Q8003
  Interventions: Drug: Low dose Q8003 (morphine sulfate and oxycodone hydrochloride)
- 3 (Active Comparator): Percocet (oxycodone and acetaminophen)
  Interventions: Drug: Percocet (oxycodone and acetaminophen)

INTERVENTIONS:
Drug: Q8003 (morphine sulfate and oxycodone hydrochloride) — IR Capsules, ascending flexible dose, every 4 to 6 hours
  Arms: 1
Drug: Low dose Q8003 (morphine sulfate and oxycodone hydrochloride) — One 3mg/2mg or 6mg/4mg IR Capsule every 4 to 6 hours
  Arms: 2
Drug: Percocet (oxycodone and acetaminophen) — One or two 5mg/325 mg tablets every 4 to 6 hours
  Arms: 3

SUMMARY:
This is a Phase 2 3-arm, open label pilot study of the safety and efficacy of Q8003 in patients who have undergone primary unilateral total knee arthroplasty or total hip arthroplasty.

DETAILED DESCRIPTION:
This Phase 2 study is a 3 arm, open-label pilot study to evaluate:

* the analgesic efficacy of a flexible ascending regimen of Q8003 compared to a low dose regimen of Q8003 (3 mg/2 mg and potentially up to 6 mg/ 4mg) and to 1-2 Percocet® 5 mg/325 mg tablets. Study drug will be administered every 4-6 hours over a 48-hour Treatment Period to inpatients with moderate to severe postoperative pain who have undergone primary unilateral total knee arthroplasty or total hip arthroplasty.
* for the flexible ascending regimen of Q8003 treatment group, to evaluate the adequacy of the algorithm for conversion of IV PCA morphine to oral morphine equivalent doses of Q8003.
* the safety of the flexible ascending regimen of Q8003 administered over a 48-hour Treatment Period.

ELIGIBILITY:
Inclusion Criteria:

* Male of female, at least 18 years of age at time of enrollment.
* If female, be at least one year post-menopausal, surgically sterile or practicing effective contraception, be non-lactating, and if of child-bearing potential, have a negative urine pregnancy test result.
* Have a body mass index (BMI) of 38 kg/m2 or less.
* Have undergone a primary unilateral total knee arthroplasty or total hip arthroplasty performed under standardized general, spinal or epidural anesthesia.
* Have developed moderate to severe pain (a score of 2 or more on the 4 point Likert scale or at least 4 on the 11 point NPRS scale within 6 hours of discontinuing PCA on the morning after surgery).

Exclusion Criteria:

* In the opinion of the Investigator, has a history of pulmonary, cardiovascular (including uncontrolled hypertension), neurologic, endocrine, hepatic, gastrointestinal, or kidney disease or therapy that, in the opinion of the Investigator, would jeopardize the patient's well being by participation in this study or is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.
* Used opiates continuously (including tramadol) for more than ten days in the past year.
* Hypersensitivity or poor tolerance to ibuprofen or short term opioids.
* Currently receiving any medications that are not at a stable dose (the same dose for > 2 months prior to date of surgery).
* Was dosed with another investigational drug within 30 days prior to the Screening Visit or has previously received treatment with Q8003.
* Current therapy with central nervous system depressant medications that might increase the risks of treatment with opioids (other than those used with surgical anesthesia).
* Current evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).
* History of abusing licit or illicit drug substances within five (5) years of study entry.
* Has taken drugs known to interact with morphine or oxycodone metabolism, including, but not limited to, phenothiazines, monoamine oxidase inhibitors (MAOI), amphetamines, and muscle relaxants within the 4 weeks prior to the date of surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Difference in pain intensity scores from baseline | 48 hours

SECONDARY OUTCOMES:
Safety: adverse events | Throughout the 48 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Patricia T. Richards, MD, Ph.D., Study Director — QRxPharma Inc.
Locations (4):
- United States (4):
  - West Alabama Research, Inc., Birmingham, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - William Beaumont Hospital, Royal Oak, Michigan
  - Research Concepts, Ltd., Houston, Texas

REFERENCES:
- [Derived] Richards P, Gimbel JS, Minkowitz HS, Kelen R, Stern W. Comparison of the efficacy and safety of dual-opioid treatment with morphine plus oxycodone versus oxycodone/acetaminophen for moderate to severe acute pain after total knee arthroplasty. Clin Ther. 2013 Apr;35(4):498-511. doi: 10.1016/j.clinthera.2013.03.002. Epub 2013 Mar 29. PMID 23545428